CLINICAL TRIAL: NCT04619095
Title: Randomised, Blinded, Parallel, Placebo-controlled Study to Evaluate Whether Supplementation of the Dietary Fiber Psyllium Can Reduce Abdominal Pain and Improve Quality of Life and Anxiety in Children With Abdominal Pain.
Brief Title: Reducing Pain and Anxiety Through Dietary Fiber Supplementation in Children With Abdominal Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to recruit any participants
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB20-1373
Record Dates: First submitted 2020-10-02; First posted 2020-11-06 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2021-09

CONDITIONS: Functional Abdominal Pain Syndrome
Keywords: Fiber; Psyllium; Quality of life; Gut microbiota; Anxiety; Pediatrics
MeSH Terms: conditions — Anxiety Disorders | interventions — Psyllium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psyllium (Experimental): For participants aged 8-11 and weighing > 24 kgs, the dosage is daily 3 grams for 2 weeks followed by daily 6 grams for 10 weeks. For children aged 12-16 and weighing > 40 kgs, the dosage is daily 5 grams for 2 weeks followed by daily 10 grams for 10 weeks.
  Interventions: Dietary Supplement: Psyllium
- Placebo (Placebo Comparator): For participants aged 8-11 and weighing > 24 kgs, the dosage is daily 3 grams for 2 weeks followed by daily 6 grams for 10 weeks. For children aged 12-16 and weighing > 40 kgs, the dosage is daily 5 grams for 2 weeks followed by daily 10 grams for 10 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Psyllium — See the information already included in the arm descriptions.
  Arms: Psyllium
Dietary Supplement: Placebo — See the information already included in the arm descriptions.
  Arms: Placebo

SUMMARY:
Background - Mental health and pain problems in early childhood are major risk factors for serious mental health problems into adulthood. These long-term effects point toward the essential need for prevention and early intervention to curbing the rising tide of global mental health disease. New approaches to child and adolescent mental health are urgently needed.

This study focus on children with functional abdominal pain (FAP), which is defined as recurrent abdominal pain independent of bowel movements without an underlying medical cause. This population has a high co-occurrence of anxiety and somatic complaints. The effects of fiber on gastrointestinal pain have not yet been tested in this group. The investigators propose that supplementation with dietary fiber (psyllium) in children with FAP will promote SCFA production by the gut microbiota, reducing abdominal pain and subsequently anxiety and improving quality of life. Psyllium promotes SCFA production, is considered safe, and meta-analyses have identified it as the most potent fiber for reducing abdominal complaints in IBS patients, indicating strong potential for reducing abdominal pain in children with FAP.

It is essential that potential mechanisms through which psyllium-induced SCFA production can reduce abdominal pain and anxiety symptoms and improve quality of life are explored. This study will explore 3 mechanisms: 1) activation of the vagus nerve, as SCFAs can induce vagal signalling, and evidence suggests that vagus nerve stimulation can reduce pain and anxiety symptoms; 2) reduction in HPA-axis responsiveness, since fiber has been shown to do so in adults, and both abdominal pain and anxiety disorders are associated with increased HPA-axis activity; and 3) structural and functional brain changes in the amygdala and hippocampus, as SCFA can influence neuronal activity of specific brain regions and probiotics-induced improvements in mental health have been related to these brain regions in adults with IBS.

Research question & Objectives - The first objective is to provide a dietary fiber psyllium supplement to children (ages 8-16 years) who suffer from FAP. The aims are to: 1) determine whether psyllium reduces abdominal pain, 2) investigate whether this subsequently decreases anxiety and improves quality of life, and 3) assess associated gut-brain axis mediators, specifically the vagus nerve, HPA-axis, and brain networks.

Methods - The investigators propose a 12-week placebo-controlled double-blind parallel-group intervention pilot study (n=20/group) where children suffering from FAP will receive a daily supplement of either psyllium or placebo (maltodextrin). For participants aged 8-11 and weighing > 24 kgs, the dosage is daily 3 grams for 2 weeks followed by daily 6 grams for 10 weeks. For children aged 12-16 and weighing > 40 kgs, the dosage is daily 5 grams for 2 weeks followed by daily 10 grams for 10 weeks. An initial lower dose was chosen to allow the gastrointestinal tract to acclimatize to the increase in dietary fiber. The dosages were chosen based on the fact that this age group typically consumes 10g less dietary fiber than recommended. All study measures are collected prior to, and after the intervention. The primary measure is abdominal pain frequency and intensity during 7 consecutive days. Secondary measures include parent and child reported anxiety and quality of life. Stool samples are used to determine gut microbiota and SCFAs. MRI will be used to assess the role of brain regions implicated in pain and anxiety. Respiratory sinus arrhythmia during seated rest will be used to assess basal vagal tone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of functional abdominal pain as defined by the Rome IV criteria for childhood functional gastrointestinal disorders

Exclusion Criteria:

* Diagnosis of inflammatory bowel disease or irritable bowel syndrome
* Lactose intolerance
* Abdominal surgery within the past year
* Contraindications for imaging
* Antibiotic use over the last 3 months

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in abdominal pain scores as measured by an abdominal pain diary | Significant change from week-zero to week 12 between the active and placebo group
  The score minimum on the scale is 0, the maximum is 20. Higher scores indicate a worse outcome.
  The abdominal pain score diary is adapted from: See et al., 2001 - DOI: 10.1023/a:1010793408132

SECONDARY OUTCOMES:
Anxiety scores as measured by PROMIS Anxiety scale | Significant change from week-zero to week 12 between the active and placebo group
  The Patient-Reported Outcomes Measurement Information System (PROMIS) questionaire will be used. The score minimum on the scale is 8, the maximum is 40. Higher scores indicate a worse outcome.
Quality of life as measured using the functional disability inventory (FDI) | Significant change from week-zero to week 12 between the active and placebo group
  The functional disability inventory (FDI) questionnaire will be used. The score minimum on the scale is 0, the maximum is 96. Higher scores indicate a worse outcome.

OTHER OUTCOMES:
Stool microbiome - Stool samples will be assayed using metagenome shotgun sequencing, after which alpha diversity is assessed. | Significant change in alpha diversity from week-zero to week 12 between the active and placebo group
  Alpha diversity will be assessed using the Shannon diversity index.
Stool metabolome - Stool samples will be assayed using liquid chromatography-mass spectrometry for short-chain fatty acid levels | Significant change in short-chain fatty acid levels from week-zero to week 12 between the active and placebo group
  Short-chain fatty acid levels are expressed as mM.
Respiratory sinus arrhythmia.This will be quantified using the high-frequency component of heart-rate variability. | Significant change from week-zero to week 12 between the active and placebo group
  Vagus nerve activity will be measured indirectly using respiratory sinus arrhythmia.
Both structural and functional MRI will be used to quantify changes in connectivity between the amygdala and prefrontal cortex. | Significant change in amygdala-prefrontal cortex connectivity from week-zero to week 12 between the active and placebo group
  Connectivity will be expressed as a z-score.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Giesbrecht, PhD, Principal Investigator — Depts. of Paediatrics and Community Health Sciences, University of Calgary
Locations (1):
- Pediatric GI Motility Laboratory at Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No